CLINICAL TRIAL: NCT06798441
Title: Determination of the Oral Irritation Potential of a Fluoride Rinse in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CS2024OC100194
Record Dates: First submitted 2025-01-14; First posted 2025-01-29 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Toothbrushing; Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brush Only (Active Comparator): All subjects will receive a marketed fluoride-containing dentifrice (Colgate® Kids Maximum Cavity Protection Pump Toothpaste) and a soft flat trimmed bristled toothbrush at their Screening/Baseline visit to use throughout the study.
  Interventions: Other: Brush Only
- Brush / Rinse (Jolly Rancher Prototype) (Experimental): All subjects will receive a marketed fluoride-containing dentifrice (Colgate® Kids Maximum Cavity Protection Pump Toothpaste) and a soft flat trimmed bristled toothbrush at their Screening/Baseline visit to use throughout the study. The subjects in this arm will receive also the assigned mouthwash (Jolly Rancher Prototype).
  Interventions: Other: Brush / Rinse (Jolly Rancher Prototype)
- Brush / Rinse (LISTERINE® Total Care Zero Alcohol) (Experimental): All subjects will receive a marketed fluoride-containing dentifrice (Colgate® Kids Maximum Cavity Protection Pump Toothpaste) and a soft flat trimmed bristled toothbrush at their Screening/Baseline visit to use throughout the study. The subjects in this arm will receive also the assigned mouthwash (LISTERINE® Total Care Zero Alcohol).
  Interventions: Other: Brush / Rinse (LISTERINE® Total Care Zero Alcohol)

INTERVENTIONS:
Other: Brush Only — Subjects will brush twice daily for one timed minute with the toothpaste and toothbrush provided. Subjects will record their twice daily product usage on a subject diary.
  Arms: Brush Only
Other: Brush / Rinse (Jolly Rancher Prototype) — Subjects will brush twice daily for one timed minute with the toothpaste and toothbrush provided. After brushing for 1 timed minute, subjects will vigorously swish with 10mL (2 teaspoons) of rinse between their teeth for 1 minute and then spit out. Subjects will record their twice daily product usage on a subject diary.
  Arms: Brush / Rinse (Jolly Rancher Prototype)
Other: Brush / Rinse (LISTERINE® Total Care Zero Alcohol) — Subjects will brush twice daily for one timed minute with the toothpaste and toothbrush provided. After brushing for 1 timed minute, subjects will vigorously swish with 10mL (2 teaspoons) of rinse between their teeth for 1 minute and then spit out. Subjects will record their twice daily product usage on a subject diary.
  Arms: Brush / Rinse (LISTERINE® Total Care Zero Alcohol)

SUMMARY:
The primary objective of this clinical trial is to determine the oral hard and soft tissue tolerance of an investigational essential oil, non-alcohol, fluoride containing mouth rinse in children 6-11 years of age compared to brushing alone and a marketed comparator mouth rinse when used as directed over a four-week period.

ELIGIBILITY:
Inclusion Criteria:

* Children, 6-11 years of age (inclusive) at the time of screening/baseline (minimum 15% Black and 5% Asian race; minimum 10% Hispanic ethnicity)
* Minimum of 16 natural teeth
* Generally, in good health
* In good oral health with adequate oral hygiene
* Willingness to participate in the clinical trial after the nature of the clinical trial has been fully explained to the child and their assent obtained
* Willingness to use the assigned products according to instructions, availability for appointments, and likelihood of completing the clinical trial
* Individual (and/or their legally acceptable representative, as applicable) has signed the Consent for Photograph Release and ICD (and/or Assent Document, as applicable) including Health Insurance Portability and Accountability Act (HIPAA) disclosure
* Absence of significant oral soft tissue pathology and active dental caries, based on the dentist's visual examination and at the discretion of the Investigator
* Able to read and understand the local language and provide written informed assent and parent/guardian to provide a signed and dated informed consent form prior to any study- related procedures

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses, and red food dye
* Use of antibiotics, or anticoagulant therapy during the study or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the investigator
* Dental prophylaxis within four weeks prior to Screening/Baseline visit
* Subjects who were previously screened and ineligible or were randomized to receive investigational product
* Significant, unstable or uncontrolled medical condition which may interfere with a subject's participation in the study, at the discretion of the Investigator
* Subjects who are related to those persons involved directly or indirectly with the conduct of this study
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e- cigarette usage
* Subjects who wear orthodontic bands, fixed retainers, removable orthodontic appliances, clear aligners or night guards or subjects who have had significant cosmetic restorations
* Hasself-reported Type 1 or Type 2 diabetes oris taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including:

  * Immunosuppressive or steroidal drugs within 2 months before Visit 1
  * Non-steroidal anti-inflammatory drugs within 5 days before Visit 1
  * Antihistamines within 2 weeks before Visit 1
* Is self-reported to be pregnant or planning to become pregnant during the study
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Participation in any clinical trial within 30 days of the Screening/Baseline visit

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Oral Tolerance as Assessed by Clinical Examinations of Oral Hard and Soft Tissues | Up to Day 28
  Oral tissue tolerance will include the assessment of the number of participants with treatment-emergent adverse events (TEAEs) and those experiencing investigational product-related AEs throughout the observational study period of 28 days. In particular, oral examinations will include clinical evaluation of soft and hard tissues, such as buccal and sublingual mucosa, tongue, hard and soft palate, gingiva, uvula, oropharynx, teeth, and dental restorations, with findings recorded in the electronic data capture (EDC) system tissues tolerance to the treatments.

SECONDARY OUTCOMES:
Parent perception questionnaire | Visit 1 (Day 0) and Visit 3 (Day 28)
  Parent perception questionnaire will be summarized at Day 0 and Day 28 by investigational product, descriptively. No statistical comparisons will be performed.
Children self-perception questionnaire | Visit 1 (Day 0) and Visit 3 (Day 28)
  Children self-perception questionnaire will be summarized at Day 0 and Day 28 by investigational product, descriptively. No statistical comparisons will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No